CLINICAL TRIAL: NCT01712997
Title: Phase Ⅲ Study of the Initial Combination of Bosentan With Iloprost in the Treatment of Pulmonary Arterial Hypertension Patients
Brief Title: Study of the Initial Combination of Bosentan With Iloprost in the Treatment of Pulmonary Hypertension Patients
Acronym: BIPH
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Air Force Military Medical University, China (Other)
Responsible Party: Principal Investigator, Shengqing Li, Associate Chief Physician, Associate Professor, Air Force Military Medical University, China
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BIPH-20121022
Record Dates: First submitted 2012-10-22; First posted 2012-10-24 (Estimated); Last update posted 2014-02-27 (Estimated); Status verified 2014-02

CONDITIONS: Pulmonary Arterial Hypertension
Keywords: Treatment of
MeSH Terms: conditions — Pulmonary Arterial Hypertension | interventions — Iloprost; Bosentan

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Combination therapy (Experimental): combine inhaled iloprost, 10μg, 4-6times/day with bosentan,125mg,po,bid.
  Interventions: Drug: Iloprost; Drug: Bosentan
- monotherapy (Active Comparator): Bosentan,125mg,po,bid.
  Interventions: Drug: Bosentan

INTERVENTIONS:
Drug: Iloprost
  Arms: Combination therapy
Drug: Bosentan

SUMMARY:
Previous studies suggest that combinations of existing therapies may be effective for pulmonary arterial hypertension (PAH). However, all of these studies are sequential combination therapy, for example, by adding sildenafil to previously prescribed bosentan. This kind of therapy model is not enough for PAH patients, especially those with New York Heart Association (NYHA) class Ⅲ and Ⅳ. In this randomized, multicenter study, the investigators evaluate the safety and efficacy of combining inhaled iloprost, a prostacyclin analog, with the endothelin receptor antagonist bosentan in treatment naive patients with PAH by comparing with bosentan monotherapy. Efficacy endpoints include change from baseline in 6-min-walk distance (6-MWD), modified (NYHA) functional class, hemodynamic parameters, and time to clinical worsening.

ELIGIBILITY:
Inclusion Criteria:

* aged 10 to 80
* treatment naive symptomatic PAH
* 6-MWD of 100-425 m
* resting mean pulmonary artery pressure greater than 25 mm Hg, pulmonary capillary wedge pressure less than 15 mm Hg, and pulmonary vascular resistance of 240 dyn.s.cm-5 or greater.

Exclusion Criteria:

* Patients with thromboembolic disease,
* untreated obstructive sleep apnea,
* portal hypertension,
* chronic liver disease or renal insufficiency,
* left-sided or unrepaired congenital heart disease,
* substantial obstructive (FEV1/FVC<50% predicted) or restrictive (total lung capacity<60% predicted) lung disease
* Patients receiving phosphodiesterase inhibitors or other prostanoids and endothelin receptor antagonists

Ages: 10 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2012-09; Primary Completion 2014-09 (Estimated)

PRIMARY OUTCOMES:
change from baseline in 6-min-walk distance (6-MWD) | 12 weeks

SECONDARY OUTCOMES:
modified (NYHA) functional class | 12 weeks

OTHER OUTCOMES:
time to clinical worsening | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Shengqing Li, MD, PhD, Principal Investigator — The department of pulmonary and critical care medicine, Xijing hospital
Locations (2):
- China (2):
  - The department of pulmonary and critical care medicine, Tangdu hospital, Xi'an, Shaanxi
  - The department of pulmonary and critical care medicine, Xijing hospital, Xi'an, Shaanxi

REFERENCES:
- [Derived] Han X, Zhang Y, Dong L, Fang L, Chai Y, Niu M, Yu Y, Liu L, Yang X, Qu S, Li S. Treatment of Pulmonary Arterial Hypertension Using Initial Combination Therapy of Bosentan and Iloprost. Respir Care. 2017 Apr;62(4):489-496. doi: 10.4187/respcare.05280. Epub 2017 Jan 24. PMID 28119496